CLINICAL TRIAL: NCT04204954
Title: A Randomized Controlled Trial of Treatment Efficacy in Ameliorating Demodex Spp. Infestation Among Cases Undergoing Cataract Surgery
Brief Title: Evaluation of Treatment Option for Demodicosis in Patients Undergoing Cataract Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital de La Luz (Other)
Collaborators: Claudia Palacio Pastrana, M.D., M.Sc. (Unknown); Samuel J. Avalos Lara, M.D. (Unknown); Hector Perez Cano, Ph.D. (Unknown); Bani Antonio-Aguirre, M.D., M.P.H.c. (Unknown); Cristina Mendoza-Velasquez, M.D., M.Sc. (Unknown); Azyadeh Camacho-Ordóñez, M.D., M.Sc.c. (Unknown); Andric C. Perez-Ortiz, M.D., M.P.H. (Unknown)
Responsible Party: Principal Investigator, Andric C Perez-Ortiz, M.D., M.P.H., Clinical Professor, Hospital de La Luz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201959B1
Record Dates: First submitted 2019-12-14; First posted 2019-12-19 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Demodex Infestation; Demodicosis; Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with Demodex spp. infestation undergoing cataract surgery were randomly allocated into four comparison groups a control group (standard treatment) and three new modalities of Demodex therapy (Blephaclean, baby shampoo, and tea tree oil) + conventional treatment.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and outcomes assessors were blinded to the treatment allocation of each participant. Outcome assessors were anterior segment surgeons who evaluated cases prior to cataract surgery. There was no indication of group allocation in the electronic medical records (EMR), only the participation of each candidate in the study. Similarly, investigators were blinded to group allocation and only recorded data directly from EMR. Blinding was kept after data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1: Topical 0.3% Ciprofloxacin [Cipro] (Other): Ciprofloxacin Ophthalmic Ointment 0.3% every four hours for three days.
  Interventions: Drug: Ciprofloxacin Ophthalmic Ointment 0.3%
- Group 2: Cipro + 50% diluted baby shampoo (Active Comparator): Ciprofloxacin Ophthalmic Ointment 0.3% every four hours for three days. Twice a day eyelid margin cleansing with 50% diluted baby shampoo for three days.
  Interventions: Drug: Ciprofloxacin Ophthalmic Ointment 0.3%; Other: Baby shampoo
- Group 3: Cipro + Blephaclean (Active Comparator): Ciprofloxacin Ophthalmic Ointment 0.3% every four hours for three days. Twice a day eyelid margin cleansing with Blephaclean Sterile Eyelid Wipes (Thea Pharmaceuticals) for three days.
  Interventions: Drug: Ciprofloxacin Ophthalmic Ointment 0.3%; Other: Blephaclean
- Group 4: Cipro + Tea tree oil. (Experimental): Ciprofloxacin Ophthalmic Ointment 0.3% every four hours for three days. Twice a day eyelid margin cleansing with tea tree oil shampoo for three days.
  Interventions: Other: Tea Tree Oil Shampoo; Drug: Ciprofloxacin Ophthalmic Ointment 0.3%

INTERVENTIONS:
Other: Tea Tree Oil Shampoo — Twice a day eyelid margin cleansing for three days.
  Arms: Group 4: Cipro + Tea tree oil.
Drug: Ciprofloxacin Ophthalmic Ointment 0.3% — Applied topically in the eyelid margin every four hours for three days.
Other: Baby shampoo — Twice a day eyelid margin cleansing for three days.
  Other Names: 50% diluted baby shampoo
  Arms: Group 2: Cipro + 50% diluted baby shampoo
Other: Blephaclean — Twice a day eyelid margin cleansing for three days.
  Arms: Group 3: Cipro + Blephaclean

SUMMARY:
Demodex blepharitis is a prevalent cause of comorbid infection among individuals undergoing cataract surgery. Several complications may arise in the postsurgical period from Staphylococcus or Streptococcus co-infections, as Demodex is a vector for these pathogens. Hence, prophylactic treatments before cataract surgery may lead to a reduction in complication rates. Since Demodex infestation and cataract surgery are two prevalent coexisting conditions in the general population, this study aims to test the effect of four combined treatments to eradicate or improve the Demodex infestation index before surgery. The investigators are conducting a single-blinded randomized trial of four therapies in participants undergoing cataract surgery. All participants will or are receiving daily eyelid cleansing bid and topical 0.3% ciprofloxacin q4h for three days added to the allocated treatment arm. Our four intervention groups are: [1] Blephaclean eye scrubs; [2] 50% dilution baby shampoo; [3] tea tree oil shampoo; [4]: topical 0.3% ciprofloxacin alone. To assess treatment efficacy, the investigators will perform eyelash hair epilation pre and postoperatively. The primary outcome is a change in the mean Demodex spp. infestation index. Also, a change in the crude number of Demodex (egg, larvae, nymph, or adult-form) spp. in eyelashes after one-week of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent after explanation of the nature and possible consequences of the study.
* Clinical diagnosis of cataracts staged with Lens Opacity Classification System III based on the American Academy of Ophthalmology and the American Society of Cataract and Refractive Surgery guidelines.
* No topical antibiotic ointment therapy or eyelid cleansing in the past six months.
* No systemic antibiotic or antiparasite treatment in the past six months.
* No ocular comorbidities (other than cataracts)
* No systemic comorbidities.

Exclusion Criteria:

* Withdrawal from the study.
* Minimal changes based on the Lens Opacity Classification System III.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Mean Demodex spp. infestation index by intervention group | One week.
  Number of demodex (egg, larvae, nymph, adult-form) spp. per eyelash (taken from epilation).
Crude count of Demodex spp. adult-forms (mites) in eyelashes by intervention group | One week.
  Number of demodex (egg, larvae, nymph, adult-form) spp. in total (taken from epilation).

SECONDARY OUTCOMES:
Endophthalmitis in the postoperative period. | One week.
  Number of cases diagnosed with endophthalmitis in the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Palacio Pastrana, M.D., M.P.H., Principal Investigator — Hospital de La Luz
Locations (1):
- Hospital de la Luz, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No